CLINICAL TRIAL: NCT07077031
Title: Comparison of Postoperative Morphine Requirements Between Two Magnesium Sulfate Administration Protocols in Opioid-Free Anesthesia for Bariatric Surgery
Brief Title: Comparison of Two Magnesium Sulfate Protocols in Opioid-Free Anesthesia for Bariatric Surgery
Acronym: OFA-MG
Status: Completed | Type: Observational
Sponsor: Hospital HM Nou Delfos (Other)
Responsible Party: Principal Investigator, HIPÓLITO LABANDEYRA GONZALEZ, Anesthesiologist, Hospital HM Nou Delfos
Other Study IDs: 25.04.2520-GHM
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain; Obesity; Bariatric Surgery; Opioid-free Anesthesia
Keywords: Magnesium Sulfate; Morphine Consumption; Opioid-Free Anesthesia; TIVA; Multimodal Analgesia
MeSH Terms: conditions — Pain, Postoperative; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TIVA-OFA Mg Bolus: Patients who received a single IV bolus of magnesium sulfate (40 mg/kg) prior to anesthesia induction, as part of an opioid-free total intravenous anesthesia (TIVA) protocol (propofol, dexmedetomidine, lidocaine, ketamine).
- TIVA-OFA Mg Bolus + Infusion: Patients who received a bolus of magnesium sulfate (50 mg/kg) followed by a continuous intraoperative infusion (15 mg/kg/h), as part of an opioid-free TIVA protocol (propofol, dexmedetomidine, lidocaine, ketamine).

SUMMARY:
This retrospective observational study aims to compare postoperative morphine consumption in patients undergoing bariatric surgery with opioid-free anesthesia (OFA) using two different intravenous magnesium sulfate administration protocols: a single bolus versus a bolus followed by continuous infusion. Medical records of 110 patients operated between June 2022 and December 2023 at Hospital HM Nou Delfos were reviewed. All patients received standardized OFA, and only the magnesium protocol varied between the groups. The primary objective was to evaluate total morphine consumption during the first 48 hours postoperatively. Secondary outcomes included pain scores, antiemetic use, and adverse events. This study was approved by the hospital's Research Ethics Committee (Protocol V3_12.05.2025).

DETAILED DESCRIPTION:
This is a retrospective, single-center, observational study conducted at Hospital HM Nou Delfos (Barcelona, Spain), which compares the effect of two intravenous magnesium sulfate (MgSO₄) administration protocols on postoperative opioid requirements in patients undergoing bariatric surgery under opioid-free anesthesia (OFA).

The two magnesium protocols evaluated were:

Group A: MgSO₄ bolus 40 mg/kg administered before induction.

Group B: MgSO₄ bolus 50 mg/kg before induction followed by continuous infusion of 15 mg/kg/h until the end of surgery.

All patients underwent standardized OFA including propofol, lidocaine, ketamine and dexmedetomidine. No intraoperative opioids were administered. Multimodal postoperative analgesia was provided in all cases(dexamethasone, paracetamol, and dexketoprofen).

A total of 110 patients were included in the analysis, as defined in the original approved protocol (55 per group).

The primary outcome was cumulative morphine consumption in the first 48 hours postoperatively.

Secondary outcomes included:

Pain scores at rest and with movement at 2, 6, 12, 24, and 48 hours

Use of rescue analgesics

Incidence of postoperative nausea and vomiting (PONV)

Adverse events potentially related to OFA (e.g., hypotension, bradycardia)

Data were extracted from electronic health records and analyzed using descriptive and inferential statistical methods. This study aims to contribute real-world evidence on magnesium strategies in OFA and to support the development of safe, cost-effective analgesic protocols in bariatric patients.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 65 years

Body mass index (BMI) ≥ 30 kg/m²

ASA physical status II or III

Underwent laparoscopic bariatric surgery (sleeve gastrectomy or Roux-en-Y gastric bypass) under opioid-free total intravenous anesthesia

Exclusion Criteria:

Pregnancy or breastfeeding

Chronic opioid use before surgery

Known allergy to magnesium sulfate or any drug used in the anesthetic protocol

Severe renal or hepatic insufficiency

Untreated coagulopathy

Active substance abuse

Uncontrolled psychiatric disorders

Intraoperative complications requiring deviation from the protocol

Postoperative morphine consumption exceeding institutional standards

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese adult patients who underwent laparoscopic bariatric surgery under opioid-free total intravenous anesthesia at a single academic center. Participants were retrospectively assigned to one of two magnesium sulfate administration protocols.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Total postoperative morphine consumption (mg) within 48 hours after surgery | 0-48 hours after surgery
  Total amount of morphine administered within 48 hours after surgery, measured in milligrams, as recorded in the post-anesthesia care unit and hospital stay.

SECONDARY OUTCOMES:
Pain intensity using Visual Analog Scale (VAS) | 1, 2, 4, 24, and 48 hours postoperatively
  Pain intensity assessed using a 10-point Visual Analog Scale (VAS), where 0 represents no pain and 10 represents the worst imaginable pain.
Incidence of adverse events | Up to 48 hours after surgery
  Number of patients experiencing side effects such as nausea, vomiting, pruritus, hypotension, bradycardia, ileus, or urinary retention.
Sleep quality reported by the patient | Within 24 hours after surgery
  Patient-reported quality of sleep using a numeric scale from 1 (very poor) to 5 (very good).
Patient satisfaction with anesthesia | Within 24 hours after surgery
  Satisfaction assessed using a standardized like scale questionnaire (1 = very dissatisfied, 5 = very satisfied).
Length of hospital stay | Up to 5 days after surgery
  Total number of days from surgery to discharge, extracted from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Contreras-Pérez, Anesthesiologist, Principal Investigator — Hospital HM Nou Delfos
Locations (1):
- Hospital HM Nou Delfos, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy regulations and ethical considerations. The dataset contains sensitive health information from a retrospective analysis and cannot be anonymized to the level required for public release. Access will be limited to the research team and authorized personnel as approved by the ethics committee.

REFERENCES:
- [Background] Alsumali A, Eguale T, Bairdain S, Samnaliev M. Cost-Effectiveness Analysis of Bariatric Surgery for Morbid Obesity. Obes Surg. 2018 Aug;28(8):2203-2214. doi: 10.1007/s11695-017-3100-0. PMID 29335933
- [Background] Schumann R. Anaesthesia for bariatric surgery. Best Pract Res Clin Anaesthesiol. 2011 Mar;25(1):83-93. doi: 10.1016/j.bpa.2010.12.006. PMID 21516916
- [Background] Shariat Moharari R, Motalebi M, Najafi A, Zamani MM, Imani F, Etezadi F, Pourfakhr P, Khajavi MR. Magnesium Can Decrease Postoperative Physiological Ileus and Postoperative Pain in Major non Laparoscopic Gastrointestinal Surgeries: A Randomized Controlled Trial. Anesth Pain Med. 2013 Dec 6;4(1):e12750. doi: 10.5812/aapm.12750. eCollection 2014 Feb. PMID 24660146
- [Background] Silva Filho SE, Dainez S, Gonzalez MAMC, Angelis F, Vieira JE, Sandes CS. Intraoperative Analgesia with Magnesium Sulfate versus Remifentanil Guided by Plethysmographic Stress Index in Post-Bariatric Dermolipectomy: A Randomized Study. Anesthesiol Res Pract. 2022 Oct 26;2022:2642488. doi: 10.1155/2022/2642488. eCollection 2022. PMID 36339775
- [Background] Levaux Ch, Bonhomme V, Dewandre PY, Brichant JF, Hans P. Effect of intra-operative magnesium sulphate on pain relief and patient comfort after major lumbar orthopaedic surgery. Anaesthesia. 2003 Feb;58(2):131-5. doi: 10.1046/j.1365-2044.2003.02999.x. PMID 12562408
- [Background] Albrecht E, Kirkham KR, Liu SS, Brull R. Peri-operative intravenous administration of magnesium sulphate and postoperative pain: a meta-analysis. Anaesthesia. 2013 Jan;68(1):79-90. doi: 10.1111/j.1365-2044.2012.07335.x. Epub 2012 Nov 1. PMID 23121612
- [Background] De Oliveira GS Jr, Castro-Alves LJ, Khan JH, McCarthy RJ. Perioperative systemic magnesium to minimize postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2013 Jul;119(1):178-90. doi: 10.1097/ALN.0b013e318297630d. PMID 23669270
- [Background] Honarmand A, Safavi M, Badiei S, Daftari-Fard N. Different doses of intravenous Magnesium sulfate on cardiovascular changes following the laryngoscopy and tracheal intubation: A double-blind randomized controlled trial. J Res Pharm Pract. 2015 Apr-Jun;4(2):79-84. doi: 10.4103/2279-042X.154365. PMID 25984545
- [Background] Hansen BA, Bruserud O. Hypomagnesemia in critically ill patients. J Intensive Care. 2018 Mar 27;6:21. doi: 10.1186/s40560-018-0291-y. eCollection 2018. PMID 29610664
- [Background] Fawcett WJ, Haxby EJ, Male DA. Magnesium: physiology and pharmacology. Br J Anaesth. 1999 Aug;83(2):302-20. doi: 10.1093/bja/83.2.302. PMID 10618948
- [Background] Murphy JD, Paskaradevan J, Eisler LL, Ouanes JP, Tomas VA, Freck EA, Wu CL. Analgesic efficacy of continuous intravenous magnesium infusion as an adjuvant to morphine for postoperative analgesia: a systematic review and meta-analysis. Middle East J Anaesthesiol. 2013 Feb;22(1):11-20. PMID 23833845
- [Background] Gozdemir M, Usta B, Demircioglu RI, Muslu B, Sert H, Karatas OF. Magnesium sulfate infusion prevents shivering during transurethral prostatectomy with spinal anesthesia: a randomized, double-blinded, controlled study. J Clin Anesth. 2010 May;22(3):184-9. doi: 10.1016/j.jclinane.2009.06.006. PMID 20400004
- [Background] Ng KT, Yap JLL, Izham IN, Teoh WY, Kwok PE, Koh WJ. The effect of intravenous magnesium on postoperative morphine consumption in noncardiac surgery: A systematic review and meta-analysis with trial sequential analysis. Eur J Anaesthesiol. 2020 Mar;37(3):212-223. doi: 10.1097/EJA.0000000000001164. PMID 31977626
- [Background] Kahraman F, Eroglu A. The effect of intravenous magnesium sulfate infusion on sensory spinal block and postoperative pain score in abdominal hysterectomy. Biomed Res Int. 2014;2014:236024. doi: 10.1155/2014/236024. Epub 2014 Mar 19. PMID 24772415
- [Background] Ahmed SA, Abdelghany MS, Afandy ME. The effect of opioid-free anesthesia on the post-operative opioid consumption in laparoscopic bariatric surgeries: A randomized controlled double-blind study. J Opioid Manag. 2022 Jan-Feb;18(1):47-56. doi: 10.5055/jom.2022.0694. PMID 35238013